CLINICAL TRIAL: NCT03211559
Title: Investigating the Effectiveness of Clinical Pilates Exercise When Applied Together With Aerobic Exercise in Patients With Ankylosing Spondylitis
Brief Title: Clinical Pilates and Aerobic Exercise in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Sevim Öksüz, Senior Instructor, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO 16/147
Record Dates: First submitted 2016-10-19; First posted 2017-07-07 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Exercise; Ankylosing Spondylitis
Keywords: ankylosing spondylitis; clinical pilates exercise; aerobic exercise; functional exercise capacity; pulmonary function
MeSH Terms: conditions — Motor Activity; Spondylitis, Ankylosing | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AEROBİC EXERCİSE (walking on treadmill) (Active Comparator): Patients walked on treadmill for 8 weeks, 3 days in a week,30-40 minutes each.
  Interventions: Other: Exercise
- Aerobic Exercise+Clinical Pilates (Experimental): Patients walked on treamill for 8 weeks, 3 days in a week, 30-40 minutes each. Additionally they did clinical pilates exercise for 8 weeks, 3 days in a week.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — clinical pilates on mat

SUMMARY:
The aim of our study is to investigate the effect of Clinical Pilates Exercises on functional status and quality of life when applied together with aerobic exercise in patients with ankylosing spondylitis (AS).

DETAILED DESCRIPTION:
According to the power analyzes 32 patients, who were diagnosed as Ankylosing spondylitis, will be taken to the study. In the first session their spinal mobility, flexibility, dynamic and static balance, back and lower limb muscle strength, pulmonary functions and pulmonary muscle strength, disease activity level, fatigue level, functional exercise capacity will be assessed to determine functional status by a physiotherapist. Also their quality of life and factors affecting the quality will be assessed. Then the patients will be divided into two exercise groups randomly. Patients in the first group will only do aerobic exercise, patients in the second group will do clinical pilates additional to the aerobic exercise which has the same protocol with the first group. Patients will do the exercise for 8 weeks, 3 times a day individually with a physiotherapist . At the end of the 8 weeks they will be assessed with the same tests again.

ELIGIBILITY:
Inclusion Criteria:

- Man and woman diagnosed with ankylosing spondylitis .

Exclusion Criteria:

* Any neurological or muscle diseases
* Inability to continuously attend the exercise program
* Visual, hearing or mental problems that could prevent communication
* Using mobility aids
* Pregnancy
* Malignity
* Having a surgery recently
* Doing exercise regularly in last 3 months.
* Having a cardiopulmonary problem which is not under control.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Aerobic capacity will be detected with submaximal exercise testing (modified Bruce protocol). | Change from Baseline and at the end of 8 weeks
  This test will be done while patients walking on TechnoGym Excitemed Treadmillde. Heart rate will be followed with polars on the chest. Medigraph V2000 device will be used to detect the oxygen amount consumed by the patient during the protocol.

SECONDARY OUTCOMES:
Lateral spinal flexion distance was measured | At the begining and at the end of 8 weeks.
  Lateral spinal flexion distance was measured with a measuring tape and recorded in centimeters.
Lumbal flexion distance was measured | At the begining and at the end of 8 weeks.
  Lumbal flexion distance was measured with a measuring tape and recorded in centimeters.
Tragus to wall distance was measured | At the begining and at the end of 8 weeks.
  Tragus to wall distance was measured with a measuring tape and recorded in centimeters.
Intermalleoler distance was measured | At the begining and at the end of 8 weeks.
  Intermalleoler distance was measured with a measuring tape and recorded in centimeters.
servical rotation was measured | At the begining and at the end of 8 weeks.
  servical rotation was measured with a goniometer and recorded in degrees.
Spinal mobility of the chest will be measured with chest circumference test. | At the begining and at the end of 8 weeks.
  Measuring tape will be placed at the 4th costa level. the circumference during deep inspiration and deep expiration will be recorded in centimeters.
Flexibility of the upper extremity will be measured with back scratch test. | At the begining and at the end of 8 weeks.
  Patients will be asked to rotate their shoulder externally with palms facing their back. Their hand fingers extend while trying to reach the lowest point the other arm internally rotates while trying to reach the highest point. Patients are asked their fingertipsto be closer to each other. If finger tips do not touch each other, the distance between them is recorded in cm assumed as a negative score, if the fingertips touch each other, then the scora is assumed as zero. If they overlap, it is recorded in cm taking as positive score. Three repetitions are performed consecutively and the best score was recorded.
Static balance of the patients will be tested with single leg stance test. | At the beginning and at the end of 6 weeks
  Performed with eyes open and arms on the hips, the participant must stand unassisted on one leg and is timed in seconds from the time one foot is flexed off the floor to the time when it touches the ground or the standing leg or an arm leaves the hips. The time passed on one leg will be recorded in seconds.
  Performed with eyes open and arms on the hips, the participant must stand unassisted on one leg and is timed in seconds from the time one foot is flexed off the floor to the time when it touches the ground or the standing leg or an arm leaves the hips. The time passed on one leg will be recorded in seconds.
Dynamic balance of the patients will be tested with functional reach test. | At the beginning and at the end of 6 weeks
  The patient is instructed to next to, but not touching, a wall and position the arm that is closer to the wall at 90 degrees of shoulder flexion with a closed fist. The assessor records the starting position at the 3rd metacarpal head on the yardstick.
  Instruct the patient to "Reach as far as you can forward without taking a step." The location of the 3rd metacarpal is recorded. Scores are determined by assessing the difference between the start and end position is the reach distance, usually measured in inches. Three trials are done and the average of the last two is noted.
Strength and endurance of the lower extremities will be tested with Chair Sit and Stand Test | At the beginning and at the end of 6 weeks
  In this test number of sitting and standing repetitions in sec. will be recorded by the physiotherapist.
The isometric strength of the back and lower extremity muscles will be measured with a dynamometer. | At the beginning and at the end of 6 weeks
  Back-D (Digital Back Muscle) dynamometer will be used to measure the strength. 3 repetitions will be done and results will be recorded in kg.
Functionality of the patients will be measured with Vath Ankylosing Spondylitis Functionality Index. | At the beginning and at the end of 6 weeks
  In that questionnaire patients will be asked to mark the best functionality level in the past week on a 10 cm- visual analogue scale.
Disease activity level be measured with Bath Ankylosing Spondylitis Disease Activity Index. | At the beginning and at the end of 6 weeks
  The BASDAI consists of a one through 10 scale (one being no problem and 10 being the worst problem) which is used to answer 6 questions pertaining to the 5 major symptoms of AS:
  Fatigue Spinal pain Joint pain / swelling Areas of localized tenderness (also called enthesitis, or inflammation of tendons and ligaments) Morning stiffness duration Morning stiffness severity
Lung volumes and pulmonary functions will be tested with spirometric function tests. | At the beginning and at the end of 6 weeks
  FUTUREMED Discovery Spirometry device will be used. Mouth piece will be placed in patients mouth. Patients will be asked to inhale and exhale 3 times. Then they will be asked to take a deep breath and exhale forcibly as quick as possible. 3 repetitions will be done and the best score will be recorded.
the strength of pulmonar muscles will be measured with Maximal Inspiratory Presssure and Maximal Expiratory Pressure inside the mouth. | At the beginning and at the end of 6 weeks
  CAREFUSİON MicroRPM device will be used to measure the pressure inside the mouth during deep inspiration and deep expiration.
Fatigue will be evaluated by the Multidimensional Fatigue Inventory (MFI) | At the beginning and at the end of 6 weeks
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. It will be filled by the patient.
Fatigue severity level of the patient will be evaluated by the Fatigue Severity Scale. | At the beginning and at the end of 6 weeks
  The Fatigue Severity Scale is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. İt will be filled by the patients.
Sleep quality level of the patient will be evaluated by the Pitsburg Sleep Quality Index . | At the beginning and at the end of 6 weeks.
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. Patient will be asked to fill this form.
Exercise capacity will be tested by the 6 minute walk test. | At the beginning and at the end of 6 weeks.
  Walked distance during 6 minutes will be recorded in meters.
Quality of life of the patients will be determined with Ankylosing Spondylitis Quality of Life Scale. | At the beginning and at the end of 6 weeks.
  The ASQoL provides a valuable tool for assessing the impact of interventions for AS and for evaluating models of service delivery. It is well accepted by patients, taking about four minutes to complete, and has excellent scaling and psychometric properties. Patients will be asked to fill the forms.
Change in the level of anxiety and depression assessed using Hospital Anxiety and Depression Scale at 6 weeks. | At the beginning and at the end of 6 weeks.
  This scale was filled by the patients. It has no special units. The elevation of the total score indicates the increased anxiety and depression levels (score out of 42).
Change in the level of fear and avoidance associated with movement assessed using the Tampa Kinesiophobia Scale at 6 weeks. | At the beginning and at the end of 6 weeks.
  This scale will be formed by the patients. If an individual receives a high score, according to the scale, this result indicates a high level of kinesiophobia. It has not a specific unit.

CONTACTS AND LOCATIONS:
Overall Officials: Oksuz, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranen University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No
Not ethical